CLINICAL TRIAL: NCT05068037
Title: Influence of Perioperative Medical Hypnosis and Acupuncture on Early Postoperative Recovery
Brief Title: Influence of Hypnoacupuncture on Early Perioperative Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Jasmina Markovic Bozic, Principal Investigator; assist. prof., MD, PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20200114
Record Dates: First submitted 2021-06-03; First posted 2021-10-05 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Postoperative Nausea and Vomiting; Acute Postoperative Pain
Keywords: MEDICAL HYPNOSIS; PERIOPERATIVE ACUPUNCTURE
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Pain, Postoperative | interventions — Acupuncture Therapy; Antiemetics

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to three arms regarding the type of intervention
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant and the outcomes assessor will not know which intervention was used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- STANDARD (Active Comparator): TCI anaesthesia with remifentanil (4-6 µg / ml) and propofol (4-6 µg / ml) Patients will receive an antiemetic (ondansetron 4 mg). The depth of anesthesia will be adjusted to maintain BIS values of 40-55. The remifentanil infusion will be adjusted according to the pain monitor values.
  Analgesia: piritramide 0.1 mg / kg and metamizole 2.5 g.
  PACU:
  Analgesia in VAS> 3: piritramide 3 mg p.p. Antiemetic for POSB: metoclopramide 10 mg
  Interventions: Other: ANTIEMETICS
- CONTROL (Active Comparator): TCI anaesthesia with remifentanil (4-6 µg / ml) and propofol (4-6 µg / ml) Group does not receive neither acupuncture nor antiemetics. The depth of anesthesia will be adjusted to maintain BIS values of 40-55. The remifentanil infusion will be adjusted according to the pain monitor values.
  Analgesia: piritramide 0.1 mg / kg and metamizole 2.5 g.
  PACU:
  Analgesia in VAS> 3: piritramide 3 mg p.p. Antiemetic for POSB: ondansetron 4 mg.
  Interventions: Other: NOTHING
- STUDY (Active Comparator): Before surgery, one of the team members will talk to the patient and perform brief medical hypnosis to gain the patient's confidence in the method and teach him the method of relaxing and building an imaginary safe place where he feels comfortable and safe. Therapeutic communication through hypnosis will be used as an additional method in order to improve the well-being and comfort of the patient, reduce stress and use sedatives.
  TCI anaesthesia with remifentanil (4-6 µg / ml) and propofol (4-6 µg / ml) Patients will receive acupuncture (PC6 and LI4 bilaterally) and no antiemetic The depth of anesthesia will be adjusted to maintain BIS values of 40-55. The remifentanil infusion will be adjusted according to the pain monitor values.
  Analgesia: piritramide 0.1 mg / kg and metamizole 2.5 g. Removal of acupuncture needles at the end of operation
  PACU:
  Analgesia in VAS> 3: piritramide 3 mg p.p. Antiemetic for POSB: ondansetron 4 mg
  Interventions: Other: ACUPUNCTURE

INTERVENTIONS:
Other: ACUPUNCTURE — standard acupuncture TCM (analgesia, vomiting)
  Arms: STUDY
Other: ANTIEMETICS — NO ACUPUNCTURE, WITH ANTIEMETICS
  Arms: STANDARD
Other: NOTHING — NO ACUPUNCTURE, NO ANTIEMETICS
  Arms: CONTROL

SUMMARY:
Perioperative stress is associated with various influences before and after surgery. Instead of benzodiazepines, patients can be calmed by non-pharmacological methods. One of these is perioperative medical hypnosis, which has also other beneficial effects such as lower opioid consumption, better wound healing, shorter hospital stays.

Acupuncture is used for analgesia. Is is effective for preventing and treating nausea and vomiting.

Hypothesis of the study is that perioperative acupuncture reduces the consumption of analgesics and anaesthetics during surgery. The investigators will also study the impact of acupuncture on postoperative nausea and vomiting and analgesic consumption in the postoperative recovery unit and the occurrence of postoperative delirium.

DETAILED DESCRIPTION:
Detailed Description: Perioperative stress is associated with the procedure itself, anaesthesia, as well as various influences before and after surgery. Patient's feeling of discomfort and anxiety in the preoperative period are treated with benzodiazepines. Although these drugs calm the patient, they are associated with the occurrence of postoperative delirium, especially in elderly patients. Instead of benzodiazepines, patients can be calmed by other non-pharmacological methods. One of these is perioperative medical hypnosis, which also has other beneficial effects such as lower opioid consumption, better wound healing, shorter hospital stays.

At the Clinical Department of Anesthesiology and Intensive Care at the University Medical Center Ljubljana, in cooperation with the Clinical Department of Neurosurgery, investigators have been routinely using perioperative medical hypnosis in awake brain surgeries since 2016 and have very good experience.

The risk of postoperative delirium is also reduced by the use of intravenous anesthesia and reduced use of opioids.

Acupuncture has been a recognized and well-established method for the treatment of acute and chronic pain by the WHO for several decades. With the right choice of points, in addition to treating pain, we can also reduce nausea and vomiting. It is a safe method in the hands of trained doctors, with virtually no side effects.

Perioperative acupuncture has a number of beneficial effects: it reduces the consumption of anesthetics and analgesics, reduces the number of perioperative complications, and protects vital organs.

With the research, investigators want to determine if acupuncture reduces the consumption of analgesics and anaesthetics during surgery. The investigators will study also the impact of acupuncture on nausea, vomiting and analgesic consumption in the postoperative recovery unit and the occurrence of postoperative delirium.

The additional value of the research will be monitoring the quality of postoperative recovery both in terms of drug consumption and recording of postoperative complications, as well as in terms of patient satisfaction and well-being.

Prevention of perioperative complications, improved quality of patient recovery and the implementation of complementary medicine methods are among the important challenges of modern, evidence-based medicine.

The prospective randomised study will include surgical patients older than 18 years, classified by the American Society of Anesthesiologists (ASA) in groups I-III, who will be scheduled for minor surgery under general anaesthesia (inguinal hernia, spine, minor plastic surgery). Patients will sign the consent for the procedure, anaesthesia and participation in the research.

Pregnant women, psychiatric patients, children, and patients who will not sign the consent or will not be capable to cooperate in the study will not be included..

Included surgeries are not a risk factor for increased nausea and vomiting. In the study group one of the team members will talk to the patient before the surgery and perform brief medical hypnosis to improve the patient's well-being and comfort.

Therefore the patient will be under less stress in the perioperative period. Prior to initiating anesthesia, patients will be randomized into three groups: patients with hypnosis and acupuncture (study), patients with antiemetic therapy (standard), patients without antiemetic and acupuncture therapy (control).The depth of anesthesia will be adjusted to maintain BIS values of 40-55. The remifentanil infusion will be adjusted according to the pain monitor values. Patients will receive analgesia according to the protocol. Investigators will collect pain and POSB data in the postoperative recovery unit and in the ward after 24 hours.

Duration of surgery and anaesthesia and the consumption of analgesics and anaesthetics will be recorded.

After three days, patients will be asked about their well-being and satisfaction.

The research will be performed by specialist anesthesiologists and an anesthesiology specialist who are trained in the pharmacological and non-pharmacological skills required for the research.

ELIGIBILITY:
Inclusion Criteria:

-Patient consent

Exclusion Criteria:

* Psychosis
* No consent for the study
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Postoperative consumption of antiemetics in mg | 24 hours
  Postoperative nausea and vomiting will be measured in mg of antiemetics in PACU

SECONDARY OUTCOMES:
Postoperative consumption of analgesics in mg | 24 hours
  Postoperative pain will be measured in mg of consumed analgetics in PACU
Degree of satisfaction | 24 hours
  Patient satisfaction will be measured in scale from 0-5, where 0 means not satisfied and 5 means very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: JASMINA MARKOVIC BOZIC, MD, PhD, Principal Investigator — UMC LJUBLJANA
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No